CLINICAL TRIAL: NCT06709469
Title: A Phase I Clinical Trial of CART Cell Therapy for Refractory/ Relapsed Acute Lymphoblastic Leukemia With Unmet Needs in Children, Adolescents and Young Adults: Feasibility and Safety Study (REALL_CART).
Brief Title: Phase I Clinical Trial of CART Cell Therapy for Refractory/Relapsed Acute Lymphoblastic Leukemia in Children, Adolescents and Young Adults
Acronym: REALL_CART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP 6614
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Phase I, open label, prospective, single center, two-armed, non-randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Children and young adults with CD19+/- CD22+ B-ALL with relapsed or refractory disease not responding to conventional chemotherapy and with no other curative therapy available.
  Interventions: Biological: Autologous CD19/CD22 CAR T cells
- Arm B (Experimental): Children and youn adults with T-ALL with relapsed or refractory disease not responding to conventional chemotherapy and with no other curative therapy available.
  Interventions: Biological: Allogeneic CART-NKG2D cells

INTERVENTIONS:
Biological: Autologous CD19/CD22 CAR T cells — A total of two doses of autologous CD19/CD22 CAR T cells (first dose of up to 0.75x106/kg fresh cells), and a second infusion of unfrozen cells (same dose) if there has been no ≥ grade 1 cytokine-release syndrome (CRS) in the next 72 h; intravenously.
  Arms: Arm A
Biological: Allogeneic CART-NKG2D cells — A total of up to 3x106/kg allogeneic CART-NKG2D cells divided in three doses of up to 1x106/kg will be infused; intravenously. First infusion of fresh cells, and the 2nd and 3rd infusion of unfrozen cells (same dose) if there has been no ≥ grade 1 CRS (every 48 hours).
  Arms: Arm B

SUMMARY:
The goal of this clinical trial is to test the feasibility and safety of an academic production of two different anti-CD19 chimeric antigen receptor T cells (CART) products according to the different biomarkers of the disease in children and young adults with relapsed/refractory CD19+ B cell acute lymphoblastic leukemia (r/r B-ALL) or relapsed/refractory T-cell acute lymphoblastic leukemia (r/r T-ALL). The main questions it aims to answer are:

1. The safety and feasibility of autologous CART-19/22 in children, adolescents and young adults with a CD19+/- CD22+ relapse/ refractory disease for a r/r B-ALL.
2. The safety and feasibility of allogeneic CART-NKG2D (chimeric-antigen receptor Natural-killer group 2, member D) in children, adolescents and young adults with r/r T-ALL.

DETAILED DESCRIPTION:
Incredible progress has been made in the treatment of relapsed/refractory CD19+ acute lymphoblastic leukemia (r/r ALL) by the application of anti-CD19 chimeric antigen receptor (CAR) T cells (CART19). However, equivalent progress has not been achieved in the treatment of relapsed/refractory T-cell acute lymphoblastic leukemia (T-ALL). Furthermore and although the majority of patients with CD19+ r/r ALL respond to CART19, 30-60% of patients relapse after this treatment, probably due to the short persistence of CAR T-cells and the immune escape or down-regulation of CD19 antigen. Patients with relapsed ALL after CART19 have a very poor prognosis and novel treatment approaches are urgently needed. To date, both relapse after CART19 malignancies and T-ALL represent an unmet medical need where no effective or targeted therapies currently exist. Recently, we and other groups have reported how T-ALL and acute myeloid leukemia (AML) cell lines were more sensitive to CART-NKG2D (chimeric-antigen receptor Natural-killer group 2, member D) cytotoxicity than B-ALL cell lines. We have previous experience in the production and administration, under compassionate use, of CART cells targeting dual CD19/CD22 antigens and NKG2D ligands. In this context, this phase I clinical trial is designed to test the feasibility and safety of an academic production of two different CART products according to the different biomarkers of the disease.

In the present study (ReALL_CART), we propose an umbrella design methodology using autologous dual CART-19/22 for CD19+/-CD22+/- relapse after CART19 or allogeneic CART-NKG2D for NKG2DL+ r/r T-ALL.

ELIGIBILITY:
Inclusion Criteria:

* ARM A: CD19+/- CD22+ B-ALL with relapsed or refractory disease not responding to conventional chemotherapy and with no other curative therapy available. Treatment with previous CART CD19 therapy is permitted, but is not mandatory, OR:
* ARM B: T-ALL with relapsed or refractory disease not responding to conventional chemotherapy and with no other curative therapy available.
* Patients diagnosed with ALL must be suitable for allogeneic HSCT and willing to proceed to transplant if the CART treatment induces complete remission and the investigator believes it is the best option.
* For ARM B there must be a suitable haploidentical donor (following local standard operating procedures).
* Lansky (age <16 years) or Karnofsky (age ≥16 years) score of 50 or greater.
* Life expectancy greater than 12 weeks.
* Absolute neutrophil count (ANC) ≥ 500/μL unless, in the opinion of the investigator, cytopenia is due to underlying leukemia and is potentially reversible with leukemia therapy.
* Platelet count ≥ 50,000/μL unless, in the opinion of the investigator, cytopenia is due to underlying leukemia and is potentially reversible with leukemia therapy.
* Absolute lymphocyte count ≥ 100/μL.
* Adequate renal, hepatic, pulmonary, and cardiac function.
* Adequate venous access and absence of contraindications for lymphoapheresis
* Patients with a seizure disorder may be enrolled if well controlled with anticonvulsants.
* Patients or patients' legal representative, parent(s), or guardian able to provide written informed consent.

Exclusion Criteria:

* Enrolled in another clinical trial in the previous 4 weeks.
* Active infection requiring systemic medical therapy including clinically significant viral infection or uncontrolled viral reactivation of EBV, CMV, adenovirus, BK-virus, HHV-6 or Aspergillus.
* Any of the following cardiac criteria: cardiac echocardiography with LVSF<30% or LVEF<40%; or clinically significant pericardial effusion.
* Presence of CNS-3 disease or uncontrolled seizure disorder.
* Active immunosuppressive therapy with the exception of prednisone 10 mg/day (or equivalent), within 7 days prior to enrolment.
* GFR <30 ml/min or bilirubin >3 times the upper limit of normality (unless due to Gilbert's syndrome).
* Any other condition that, in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the trial.
* Pregnant or lactating women.
* Sexually active patients must be willing to utilize one of the more effective birth control methods for at least 12 months after the infusion and until CAR-T cells are no longer present on two consecutive tests. Male partner should use a condom. Women of child-bearing potential are defined as all women physiologically capable of becoming pregnant.
* Sexually active males should use a condom during intercourse for at least 12 months after the infusion and until CAR-T cells are no longer present on two consecutive tests.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events in patients that received autologous CART-19/22 | Through study completion, an average of 5 years
  An adverse event is any harmful and unintended reaction to an investigational medicinal product, regardless of the dose administered.
  Adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with the exception of CRS and ICANS, which will be graded according to ASBMT Consensus Grading. If CTCAE grading does not exist for an AE, the severity of mild, moderate, severe, life-threatening and fatal, corresponding to Grades 1-5, will be used.
Incidence and severity of adverse events in patients that received allogenic CART-NKG2D T | Through study completion, an average of 5 years
  An adverse event is any harmful and unintended reaction to an investigational medicinal product, regardless of the dose administered.
  Adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with the exception of CRS and ICANS, which will be graded according to ASBMT Consensus Grading. If CTCAE grading does not exist for an AE, the severity of mild, moderate, severe, life-threatening and fatal, corresponding to Grades 1-5, will be used.

SECONDARY OUTCOMES:
Expression of CD19/CD22 and NKG2DL on primary B- or T- cell ALL, respectively | Through study completion, an average of 5 years
  The expression of CD19/CD22 and NKG2DL on primary B and T cell malignancies will be measured, respectively, by flow cytometry.
Persistence of CART19/22 and CART-NKG2D cells in patients' samples | Through study completion, an average of 5 years
  The persistance of CART19/22 and CART-NKG2D cells in patients' blood, bone marrow and cerebrospinal fluid samples will be measured
Cytokine profile | Through study completion, an average of 5 years
  Peripheral blood cytokine profile from the patients' serum. The following cytokines will be analysed: IFN-γ, TNF-α, GMCSF, IL-2, IL-1ß, IL-6, IL-8, IL-10, IL12
DNA methylation profile of NKG2DL | Through study completion, an average of 5 years
  Identify the DNA methylation profile of NKG2DL (MICA, MICB AND ULBPs 1-3) in primary T-cell malignancies' samples. This outcome will only be measured in arm B.
Presence of soluble NKG2DL, and ANTI-MICA and ANTI-MICB antibodies | Through study completion, an average of 5 years
  Evaluate the presence of soluble NKG2DL and ANTI-MICA and ANTI-MICB antibodies in the serum of patients under CART-NKG2D therapy. This outcome will only be measured in arm B.
Overall rate response in both arms | Through study completion, an average of 5 years
  Response assessment will be measured by bone marrow aspirate (or trephine in case of dry tap).

OTHER OUTCOMES:
Incidence of serious adverse events | Through study completion, an average of 5 years
  Serious adverse events are described as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly or birth defect
  * Other important medical events
Performance status | Through study completion, an average of 5 years
  The performance status of the included patients will be measured by the Lansky scale if they are younger than 16 years old, or by the Karnofsky scale if they are 16 years old or older.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Martinez B, Galan-Gomez V, Navarro-Zapata A, Mirones-Aguilar I, Cobo M, Pernas-Sanchez A, Vallejo S, Sanchez-Zapardiel E, Leon-Triana O, Echecopar C, Martinez-Romera I, Guerra-Garcia P, San Roman-Pacheco S, Escudero A, Izquierdo E, Izquierdo M, Naharro S, Martin-Ayuso A, Bareke H, Paris-Munoz A, Hu P, Schneider D, Orentas RJ, Minguillon J, Perez-Martinez A. Tandem CD19/CD22 CAR T-cells as potential therapy for children and young adults with high-risk r/r B-ALL. EBioMedicine. 2025 Aug;118:105872. doi: 10.1016/j.ebiom.2025.105872. Epub 2025 Aug 5. PMID 40753722